CLINICAL TRIAL: NCT04751396
Title: Testing of an Educational Tool for Patients With Melanoma and Concomitant Autoimmune Disease Who Are Candidates for Adjuvant Therapy With Immune Checkpoint Inhibitors: Acceptability and Usability With Patients and Providers
Brief Title: Testing of an Educational Tool for Patients With Melanoma and Pre-Existing Autoimmune Disease Who Are Candidates for Immune Checkpoint Inhibitors
Status: Recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2020-0843; NCI-2021-00565 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0843 (Other: M D Anderson Cancer Center); K08CA237619 (NIH)
Record Dates: First submitted 2021-02-08; First posted 2021-02-12 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Ankylosing Spondylitis; Autoimmune Disease; Crohn Disease; Enteropathic Arthritis; Enteropathic Spondylitis; Inflammatory Bowel Disease; Melanoma; Psoriasis; Psoriatic Arthritis; Reactive Arthritis; Rheumatoid Arthritis; Systemic Lupus Erythematosus; Ulcerative Colitis
MeSH Terms: conditions — Spondylitis, Ankylosing; Autoimmune Diseases; Crohn Disease; Inflammatory Bowel Diseases; Melanoma; Psoriasis; Arthritis, Psoriatic; Arthritis, Reactive; Arthritis, Rheumatoid; Lupus Erythematosus, Systemic; Colitis, Ulcerative | interventions — Practice Guidelines as Topic; Standard of Care; Early Intervention, Educational; Educational Status; Methods; Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Part A (Interview): Participants navigate the educational tool over 30-45 minutes then participate in an interview about their thoughts and opinions about the content, ease of use, and format of the tool over 45 minutes.
  Interventions: Other: Educational Intervention; Other: Interview
- Part B Group I (standard information): Patients receive standard educational information during their clinician encounter. Patients also complete questionnaires over 30-45 minutes at baseline within a week prior to their clinician encounter, immediately after the encounter, and at 3 months.
  Interventions: Other: Best Practice; Other: Questionnaire Administration; Other: Survey Administration
- Part B Group II (educational tool): Patients navigate educational tool over 20 minutes during their clinician encounter. Patients also complete questionnaires over 30-45 minutes at baseline within a week prior to their clinician encounter, immediately after the encounter, and at 3 months.
  Interventions: Other: Educational Intervention; Other: Questionnaire Administration; Other: Survey Administration

INTERVENTIONS:
Other: Best Practice — Receive standard educational information
  Other Names: standard of care; standard therapy
  Groups: Part B Group I (standard information)
Other: Educational Intervention — Navigate educational tool
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
  Groups: Part A (Interview); Part B Group II (educational tool)
Other: Interview — Participate in interview
  Groups: Part A (Interview)
Other: Questionnaire Administration — Complete questionnaire
  Groups: Part B Group I (standard information); Part B Group II (educational tool)
Other: Survey Administration — Complete surveys
  Groups: Part B Group I (standard information); Part B Group II (educational tool)

SUMMARY:
This study learn how easily patients can use an educational tool that will be created for patients with melanoma and pre-existing autoimmune diseases who receive or will receive immune checkpoint inhibitor drugs. Patients will be asked their opinions about the design, accessibility, and content of the tool. Researchers will use the information collected to improve the educational materials that will help patients make future decisions about their treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the acceptability (e.g., ease of use, design, accessibility, content) of the educational tool that will be developed for patients with melanoma and pre-existing autoimmune conditions considering or undergoing treatment with immune checkpoint inhibitors.

II. To test the usability in real world-settings of the educational tool (to be developed) and evaluate feasibility of patient recruitment (i.e., ability to identify enough patients and consent at least 50% of the identified patients) in a pilot study.

OUTLINE:

PART A: Participants navigate the educational tool over 30-45 minutes then participate in an interview about their thoughts and opinions about the content, ease of use, and format of the tool over 45 minutes.

PART B: 2 group of participants will be evaluated sequentially (Participants in group II will be enrolled after all the participants in group I have been assessed).

GROUP I: Patients receive standard educational information during their clinician encounter. Patients also complete questionnaires over 30-45 minutes at baseline within a week prior to their clinician encounter, immediately after the encounter, and at 3 months.

GROUP II: Patients navigate educational tool over 20 minutes during their clinician encounter. Patients also complete questionnaires over 30-45 minutes at baseline within a week prior to their clinician encounter, immediately after the encounter, and at 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of melanoma
* Diagnosis of pre-existing autoimmune disease

  * Inflammatory bowel disease

    * Diagnosis of Crohn's disease or ulcerative colitis by a gastroenterologist
    * For ulcerative colitis, proof of chronic changes over time (i.e., 6 months) and signs of inflammation histologically
    * Treatment with aminosalicylates, corticosteroids, thiopurines, or immune modifiers (e.g., calcineurin inhibitors, methotrexate, adhesion molecule antagonists)
  * Rheumatoid arthritis

    * Diagnosis of rheumatoid arthritis by a rheumatologist
    * Treatment with traditional disease-modifying antirheumatic drugs (e.g., methotrexate, sulfasalazine, hydroxychloroquine) or targeted therapy
  * Systemic lupus erythematosus

    * Diagnosis of systemic lupus erythematosus by a rheumatologist
  * Psoriasis

    * Diagnosis of psoriasis by a dermatologist
    * Treatment with corticosteroids, vitamin D analogs, anthralin, topical retinoids, calcineurin inhibitors, salicylic acid, coal tar, or moisturizers; light therapy, including sunlight, ultraviolet B (UVB) phototherapy, narrowband UVB therapy, Goeckerman therapy, photochemotherapy, excimer laser, or pulsed dye laser; or systemic medications, including retinoids, methotrexate, cyclosporine, hydroxyurea, or thioguanine or targeted therapies
  * Spondyloarthropathies

    * Diagnosis of ankylosing spondylitis, reactive arthritis, psoriatic arthritis, or enteropathic arthritis/spondylitis by a rheumatologist
    * Treatment with disease-modifying antirheumatic drugs (e.g., sulfasalazine) or targeted therapy
* Age of 18 years or older
* Patients whose physicians had recommended they begin using any of the currently available immune checkpoint inhibitors or people who are in the midst of or have already made the decision on whether or not start an immune checkpoint inhibitor
* E-mail access and computer with Internet access or telephone
* Ability to communicate in English or Spanish
* CLINICIAN
* Prescribed immune checkpoint inhibitors
* Are providing care for patients with melanoma
* In the clinics at MD Anderson

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with melanoma or pre-existing autoimmune disease and clinicians
Sampling Method: Non-Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2022-04-20 (Actual); Primary Completion 2027-02-02 (Estimated); Study Completion 2027-02-02 (Estimated)

PRIMARY OUTCOMES:
Decisional conflict scale | Up to 4 years
  The scale will be used to assess personal perceptions of 1) uncertainty in choosing among options; 2) modifiable factors contributing to uncertainty, such as feeling uninformed, and 3) feeling that the choice is values-based and likely to be implemented.

SECONDARY OUTCOMES:
Knowledge | Up to 3 months
  Will be assessed using a questionnaire developed by the research team covering various content areas, including general information about immune checkpoint inhibitors and the associated adverse effects and benefits of the treatments.
Acceptability | Immediately after the clinical encounter
  A standard assessment questionnaire will be used to obtain users' ratings of various features of the educational tool, including ease of use, presentation, usefulness and satisfaction. The items in the questionnaire come from the Ottawa Acceptability Measures.
Usability | Immediately after the clinical encounter
  A standard assessment questionnaire will be used to obtain users' ratings of various features of the educational tool, including ease of use, presentation, usefulness and satisfaction. The items in the questionnaire come from the Ottawa Acceptability Measures.
Depression | Up to 3 months
  Will be assessed using the Depression and Anxiety Stress Scale (DASS). The DASS is a 21-item self report instrument designed to measure the three related negative emotional states of depression, anxiety and tension/stress. The Depression scale assesses dysphoria, hopelessness, devaluation of life, self-deprecation, lack of interest/involvement, anhedonia, and inertia
Anxiety | Up to 3 months
  Will be assessed using the DASS. The DASS is a 21-item self report instrument designed to measure the three related negative emotional states of depression, anxiety and tension/stress. The Anxiety scale assesses autonomic arousal, skeletal muscle effects, situational anxiety, and subjective experience of anxious affect.
Stress | Up to 3 months
  Will be assessed using the DASS. The DASS is a 21-item self report instrument designed to measure the three related negative emotional states of depression, anxiety and tension/stress. The Stress scale is sensitive to levels of chronic non-specific arousal. It assesses difficulty relaxing, nervous arousal, and being easily upset/agitated, irritable/over-reactive and impatient.
CollaboRATE measure | Immediately after the clinical encounter
  The CollaboRATE questions ask about the effort made to help patients understand their health issues, listen to what matters most to them, and include what matters most to them in choosing what to do next.
Shared decision-making process survey | Immediately after the clinical encounter
  This instrument measures the extent to which health care providers engage patients in shared decision making. Items are focused on four specific behaviors that are critical for shared decision making -discussion of options, pros, cons and preferences.
Patient's perception of usefulness of the tool | Immediately after the clinical encounter
  Will use the Preparation for Decision Making Scale (Prep-DM) to assess the patients' perception of how useful the educational tool is in preparing them to communicate with their practitioner at a consultation. It is a 10-item scale developed to evaluate decision processes relating to the preparation of patients for decision making and dialoguing with their practitioners.

CONTACTS AND LOCATIONS:
Overall Officials: Angeles Lopez-Olivo, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org